CLINICAL TRIAL: NCT00693056
Title: A Double-Blinded, Randomized, Placebo-Controlled, Dose-Exploring Study of RX-10100 for Eight Weeks of On-Demand Administration in Subjects With Erectile Dysfunction (ED)
Brief Title: Efficacy Study of RX-10100 to Treat Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rexahn Pharmaceuticals, Inc. (Industry)
Responsible Party: Hyungjoo Lee / Associate Director, Product Development Management, Rexahn Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RX-10100-P2A-001
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Erectile Dysfunction (ED)
Keywords: Erectile Dysfunctions; ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — RX-10100

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: RX-10100 5mg
- 3 (Experimental)
  Interventions: Drug: RX-10100 10mg
- 4 (Experimental)
  Interventions: Drug: RX-10100 15mg

INTERVENTIONS:
Drug: Placebo — Placebo (w/o API)
  Arms: 1
Drug: RX-10100 5mg — 5 mg/dose of RX-10100
  Other Names: Zoraxel
  Arms: 2
Drug: RX-10100 10mg — 10 mg/dose of RX-10100
  Other Names: Zoraxel
  Arms: 3
Drug: RX-10100 15mg — 15 mg/dose of RX-10100
  Other Names: Zoraxel
  Arms: 4

SUMMARY:
The primary objective of this Phase IIa trial is to determine the effective doses and treatment period for an upcoming RX-10100 Phase IIb trial in subjects with erectile dysfunction (ED). The secondary objectives of this trial are to evaluate the safety and the quality of life in subjects with ED receiving RX-10100 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have had ED for at least six months
* Stable, heterosexual relationship for at least 3 months
* Make at least one attempt of sexual intercourse per week during the untreated, 2-week screening period
* At least 50% of attempts of sexual intercourse during the untreated baseline period must be unsuccessful
* 'Moderate' or 'mild to moderate' ED, defined as an IIEF-EF domain score between 11 and 21 measured

Exclusion Criteria:

* Following previous or current medical conditions

  * Any unstable medical, psychiatric, or substance abuse disorder
  * Penile anatomical abnormalities
  * Primary hypoactive sexual desire
  * Spinal cord injury
  * Hypogonadism
  * Surgical prostatectomy
  * Stable or unstable angina pectoris
  * Myocardial infarction, stroke, or life-threatening arrhythmia
  * Uncontrolled atrial fibrillation/flutter at screening
  * Severe chronic or acute liver disease
  * Moderate or severe hepatic impairment
  * Clinically significant chronic hematological disease
  * Bleeding disorder
  * Significant active peptic ulcer disease
  * Resting hypotension or hypertension
  * Malignancy (cancers)
  * NYHA Class II to IV heart failures
  * Positive test for Hepatitis B surface antigen (HBsAg) or Hepatitis C
  * Symptomatic postural hypotension
* Following concomitant medication

  * Androgens or estrogens
  * Anti-androgens
  * Potent inhibitors of cytochrome P450 3A4
  * Any other investigational drug within 30 days before Visit 1
  * Any treatment for ED within 7 days before Visit 1 or during the study
  * Antibiotics in the penicillin class
* Following abnormal laboratory values

  * Serum total testosterone level (at least 25% lower)
  * Serum creatinine (> 3.0 mg/dl)
  * Elevation of AST and/or ALT (> 3 times the upper limit of normal)
  * Diabetic subjects with an HbAlc (> 6.5%)
* Subjects with known hypersensitivity to amoxicillin
* Subjects with a history of unresponsiveness to any PDE5 Inhibitor treatment or a history of significant side effects leading to its treatment discontinuation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Scores on IIEF-EF Questionnaires and on SEP Questions II and III | Weeks 4 and 8

SECONDARY OUTCOMES:
Scores on other domains of IIEF, other questions on Subject Diaries, RigiScan measurement, and ED-QoL questionnaires | Weeks 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Hyungjoo Hugh Lee, MS, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Greenbelt, Maryland
  - Woodlane, New Jersey
  - Greer, South Carolina